CLINICAL TRIAL: NCT07221149
Title: ROSETTA Gastric-204: A Blinded, Randomized, Phase 2/3 Study of Pumitamig in Combination With Chemotherapy Versus Nivolumab in Combination With Chemotherapy in Participants With Previously Untreated Advanced or Metastatic Gastric, Gastroesophageal Junction, or Esophageal Adenocarcinoma
Brief Title: A Study to Evaluate the Safety and Efficacy of Pumitamig in Combination With Chemotherapy Versus Nivolumab in Combination With Chemotherapy in Participants With Previously Untreated Advanced or Metastatic Gastric, Gastroesophageal Junction, or Esophageal Adenocarcinoma (ROSETTA Gastric-204)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA266-0004; 2025-523263-37 (Other: EU CTR); U1111-1325-8116 (Other: WHO)
Record Dates: First submitted 2025-10-23; First posted 2025-10-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Untreated Advanced or Metastatic Gastric, Gastroesophageal Junction, or Esophageal Adenocarcinoma
Keywords: Gastric Cancer; Gastroesophageal Junction Cancer; Esophageal Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Folfox protocol; Nivolumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A1 (Experimental)
  Interventions: Drug: Pumitamig; Drug: Folfox
- Arm A2 (Experimental)
  Interventions: Drug: Pumitamig; Drug: Folfox
- Arm B (Experimental)
  Interventions: Drug: Folfox; Drug: Nivolumab
- Arm C (Experimental)
  Interventions: Drug: Pumitamig; Drug: Folfox; Drug: Capox
- Arm D (Experimental)
  Interventions: Drug: Folfox; Drug: Capox; Drug: Nivolumab

INTERVENTIONS:
Drug: Pumitamig — Specified dose on specified days
  Other Names: BMS-986545; BNT327; PM8002
  Arms: Arm A1; Arm A2; Arm C
Drug: Folfox — Specified dose on specified days
Drug: Capox — Specified dose on specified days
  Arms: Arm C; Arm D
Drug: Nivolumab — Specified dose on specified days
  Arms: Arm B; Arm D

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Pumitamig in combination with chemotherapy versus Nivolumab in combination with chemotherapy in participants with previously untreated advanced or metastatic gastric, gastroesophageal junction, or esophageal adenocarcinoma

ELIGIBILITY:
Inclusion Criteria

* Participants must be previously untreated with systemic treatment for advanced/metastatic disease, histologically or cytologically confirmed advanced or metastatic gastric cancer (GC), gastroesophageal junction adenocarcinoma (GEJC) or distal esophageal adenocarcinoma (EAC). GEJ involvement can be confirmed via biopsy, endoscopy, or imaging.
* Participants must have a documented programmed cell death-(ligand)1 (PD-L1) ≥ 1.
* Participants must have documented human epidermal growth factor receptor 2 (HER2)-negative cancer, as determined according to local guidelines.
* Participants must have measurable disease as defined by RECIST v1.1.

Exclusion Criteria

* Participants must not have untreated known central nervous system (CNS) metastases.
* Participants must not have significant cardiovascular disease, such as myocardial infarction, unstable angina, arterial thrombosis, cerebrovascular accident within 6 months prior to randomization, uncontrolled hypertension (≥ 160 systolic, ≥ 100 diastolic mm Hg) despite optimal medical management, or congenital long QT syndrome.
* Participants must not have evidence of major coagulation disorders (eg, hemophilia).
* Participants must not have a history of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism within 3 months prior to randomization, unless the participant has been fully treated (eg, inferior vena cava filter placed) and/or adequately anticoagulated on a prophylactic dose.
* Participants must not have a history of abdominal fistula or gastrointestinal (GI) perforation within 6 months of randomization.
* Participants must not have had major surgery, open biopsy, or significant traumatic injury within 28 days prior to randomization, or anticipation of the need for major surgery during the course of study intervention.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2030-11-08 (Estimated); Study Completion 2032-09-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response (OR) (confirmed complete response (CR) or partial response (PR)) by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 per investigator assessment | Up to 2 years after the last participant is randomized
  Phase 2
Progression Free Survival (PFS) by RECIST v1.1 per blinded independent central review (BICR) | Up to approximately 33 months
  Phase 3
Overall survival (OS) | Up to approximately 47 months
  Phase 3

SECONDARY OUTCOMES:
PFS by RECIST v1.1 per investigator assessment | Up to approximately 33 months
  Phase 2
Duration of Response (DOR) (CR or PR) by RECIST v1.1 per investigator assessment | Up to approximately 33 months
  Phase 2
Time to Response (TTR) (CR or PR) by RECIST v1.1 per investigator assessment | Up to approximately 33 months
  Phase 2
Disease control (Best Overall Response (BOR) of confirmed CR, confirmed PR, or Stable Disease (SD)) by RECIST v1.1 per investigator assessment | Up to approximately 33 months
  Phase 2
Recommended dose of Pumitamig for Phase 3 | Up to approximately 33 months
  Phase 2
Objective response (OR) by RECIST v1.1 per BICR | Up to approximately 33 months
  Phase 3
DOR by RECIST v1.1 per BICR | Up to approximately 33 months
  Phase 3

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (161):
- United States (32):
  - Local Institution - 0284, Phoenix, Arizona
  - Local Institution - 0240, Los Angeles, California
  - Local Institution - 0277, Orange, California
  - Local Institution - 0428, San Francisco, California
  - Local Institution - 0429, Fort Myers, Florida
  - Local Institution - 0433, Jacksonville, Florida
  - Local Institution - 0430, St. Petersburg, Florida
  - Local Institution - 0246, Tampa, Florida
  - Local Institution - 0377, Atlanta, Georgia
  - Local Institution - 0379, Chicago, Illinois
  - Local Institution - 0268, Iowa City, Iowa
  - Local Institution - 0259, Rochester, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Local Institution - 0286, Omaha, Nebraska
  - Local Institution - 0386, Lake Success, New York
  - Local Institution - 0242, New York, New York
  - Local Institution - 0274, Rochester, New York
  - Local Institution - 0222, Cleveland, Ohio
  - Local Institution - 0432, Eugene, Oregon
  - Local Institution - 0419, Portland, Oregon
  - Local Institution - 0407, Pittsburgh, Pennsylvania
  - Local Institution - 0255, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Local Institution - 0423, Amarillo, Texas
  - Texas Oncology-Austin Central, Austin, Texas
  - Local Institution - 0424, Beaumont, Texas
  - Local Institution - 0415, Denison, Texas
  - Local Institution - 0421, Grapevine, Texas
  - Local Institution - 0233, Houston, Texas
  - Local Institution - 0427, San Antonio, Texas
  - Local Institution - 0413, Salem, Virginia
  - Local Institution - 0271, Madison, Wisconsin
- Argentina (4):
  - Local Institution - 0061, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0066, ABB, Buenos Aires F.D.
  - Local Institution - 0069, Buenos Aires
  - Local Institution - 0054, Buenos Aires
- Australia (5):
  - Local Institution - 0080, Birtinya, Queensland
  - Local Institution - 0077, Elizabeth Vale, South Australia
  - Local Institution - 0085, Clayton, Victoria
  - Local Institution - 0400, Melbourne, Victoria
  - Local Institution - 0083, Perth, Western Australia
- Brazil (6):
  - Local Institution - 0208, Fortaleza, Ceará
  - Local Institution - 0204, Belo Horizonte, Minas Gerais
  - Local Institution - 0226, Natal/RN, Rio Grande do Norte
  - Local Institution - 0210, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0425, Santa Maria, Rio Grande do Sul
  - Local Institution - 0221, São José do Rio Preto
- Canada (4):
  - Local Institution - 0088, Calgary, Alberta
  - Local Institution - 0119, Halifax, Nova Scotia
  - Local Institution - 0121, Toronto, Ontario
  - Local Institution - 0175, Sherbrooke, Quebec
- Chile (3):
  - Local Institution - 0068, Santiago, Santiago Metropolitan
  - Local Institution - 0056, Santiago, Santiago Metropolitan
  - Local Institution - 0055, Santiago, Santiago Metropolitan
- China (24):
  - Local Institution - 0410, Beijing, Beijing Municipality
  - Local Institution - 0418, Beijing, Beijing Municipality
  - Local Institution - 0276, Fuzhou, Fujian
  - Local Institution - 0232, Guangzhou, Guangdong
  - Local Institution - 0280, Guangzhou, Guangdong
  - Local Institution - 0231, Nanning, Guangxi
  - Local Institution - 0237, Harbin, Heilongjiang
  - Local Institution - 0282, Weihui, Henan
  - Local Institution - 0249, Zhengzhou, Henan
  - Local Institution - 0412, Wuhan, Hubei
  - Local Institution - 0279, Wuhan, Hubei
  - Local Institution - 0292, Changsha, Hunan
  - Local Institution - 0409, Nanchang, Jiangxi
  - Local Institution - 0244, Shenyang, Liaoning
  - Local Institution - 0239, Xi'an, Shaanxi
  - Local Institution - 0266, Xi'an, Shaanxi
  - Local Institution - 0273, Jinan, Shandong
  - Local Institution - 0258, Shanghai, Shanghai Municipality
  - Local Institution - 0243, Taiyuan, Shanxi
  - Local Institution - 0260, Chengdu, Sichuan
  - Local Institution - 0248, Tianjin, Tianjin Municipality
  - Local Institution - 0408, Hangzhou, Zhejiang
  - Local Institution - 0252, Hangzhou, Zhejiang
  - Local Institution - 0269, Shanghai
- Colombia (2):
  - Local Institution - 0399, Pasto, Departamento de Nariño
  - Local Institution - 0398, Cali, Valle del Cauca Department
- France (7):
  - Local Institution - 0064, Brest, Finistère
  - Local Institution - 0062, Nantes, Pays de la Loire Region
  - Local Institution - 0051, Lille
  - Local Institution - 0058, Lyon
  - Local Institution - 0060, Marseille
  - Local Institution - 0049, Paris
  - Local Institution - 0046, Poitiers
- Germany (8):
  - Local Institution - 0089, Berlin
  - Local Institution - 0134, Frankfurt
  - Local Institution - 0090, Hamburg
  - Local Institution - 0100, Heidelberg
  - Local Institution - 0112, Leipzig
  - Local Institution - 0105, Mainz
  - Local Institution - 0101, Mannheim
  - Local Institution - 0117, Ulm
- India (7):
  - Local Institution - 0306, Nashik, Dādra and Nagar Haveli and Damān and Diu
  - Local Institution - 0305, Mumbai, Maharashtra
  - Local Institution - 0404, Mumbai, Maharashtra
  - Local Institution - 0303, Delhi
  - Local Institution - 0403, Delhi
  - Local Institution - 0302, Puducherry
  - Local Institution - 0310, Pune
- Italy (6):
  - Local Institution - 0167, Napoli, Campania
  - Local Institution - 0166, Turin, Piedmont
  - Local Institution - 0171, Milan
  - Local Institution - 0163, Milan
  - Local Institution - 0168, Padua
  - Local Institution - 0170, Roma
- Japan (15):
  - Local Institution - 0014, Chiba, Chiba
  - Local Institution - 0012, Matsuyama, Ehime
  - Local Institution - 0029, Kurashiki, Okayama-ken
  - Local Institution - 0004, Osaka, Osaka
  - Local Institution - 0028, Suita, Osaka
  - Local Institution - 0376, Takatsuki, Osaka
  - Local Institution - 0026, Nagaizumi-cho,Sunto-gun, Shizuoka
  - Local Institution - 0003, Chuo-ku, Tokyo
  - Local Institution - 0008, Koto-ku, Tokyo
  - Local Institution - 0013, Chikusa-ku
  - Local Institution - 0006, Gifu
  - Local Institution - 0033, Kashiwa
  - Local Institution - 0002, Minami-Ku, Fukuoka
  - Local Institution - 0024, Sendai
  - Local Institution - 0015, Yokohama
- Mexico (4):
  - Local Institution - 0396, Mexico City, DIF
  - Local Institution - 0395, Mexico City, Mexico City
  - Local Institution - 0397, Mexico City, Mexico City
  - Local Institution - 0394, Oaxaca City, Oaxaca
- Poland (5):
  - Local Institution - 0336, Jelenia Góra, Lower Silesian Voivodeship
  - Local Institution - 0339, Wieliszew, Masovian Voivodeship
  - Local Institution - 0342, Krakow
  - Local Institution - 0361, Krakow
  - Local Institution - 0320, Opole
- Romania (6):
  - Local Institution - 0010, Cluj-Napoca, Cluj
  - Local Institution - 0019, Cluj-Napoca
  - Local Institution - 0011, Craiova
  - Local Institution - 0030, Floresti/ Cluj
  - Local Institution - 0021, Iași
  - Local Institution - 0005, Iași
- South Korea (5):
  - Local Institution - 0034, Seongnam, Kyǒnggi-do
  - Local Institution - 0027, Seoul, Seoul Teugbyeolsi
  - Local Institution - 0020, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0001, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0036, Seoul, Seoul-teukbyeolsi
- Spain (7):
  - Local Institution - 0350, Santander, Cantabria
  - Local Institution - 0391, Pamplona, Navarre
  - Local Institution - 0312, Valencia, Valenciana, Comunitat
  - Local Institution - 0389, Madrid
  - Local Institution - 0358, Madrid
  - Local Institution - 0360, Madrid
  - Local Institution - 0390, Málaga
- Turkey (Türkiye) (5):
  - Local Institution - 0111, Ankara
  - Local Institution - 0108, Edirne
  - Local Institution - 0125, Kadiköy/Istanbul
  - Local Institution - 0093, Manisa
  - Local Institution - 0128, Sakarya
- United Kingdom (6):
  - Local Institution - 0176, Southampton, Hampshire
  - Local Institution - 0331, Manchester, Lancashire
  - Local Institution - 0316, London, London, City of
  - Local Institution - 0317, Oxford, Oxfordshire
  - Local Institution - 0354, Glasgow
  - Local Institution - 0357, Sutton

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07221149.html